CLINICAL TRIAL: NCT00471406
Title: Photodynamic Therapy With Verteporfin for Corneal Neovascularization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chonnam National University Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CPDT-0001
Record Dates: First submitted 2007-05-08; First posted 2007-05-09 (Estimated); Last update posted 2008-10-17 (Estimated); Status verified 2008-10

CONDITIONS: Corneal Neovascularization
MeSH Terms: conditions — Corneal Neovascularization | interventions — Photochemotherapy; Verteporfin

INTERVENTIONS:
Procedure: Photodynamic Therapy with Verteporfin

SUMMARY:
Purpose: To investigate the efficacy of photodynamic therapy with verteporfin for the treatment of patients with corneal neovascularization.

Design: Prospective, non-comparative case series. Participants: Eighteen eyes of 18 patients with stable corneal neovascularization who were refractory to conventional treatment.

Methods: The patients were treated with photodynamic therapy with verteporfin (6 mg/m2). Five patients were treated following penetrating keratoplasty, and 2 patients were treated before penetrating keratoplasty. Best corrected visual acuity and anterior segment photography were performed before and after treatment. The length of cumulative blood vessels and area of corneal neovascularization were measured.

Main outcome measures: Vascular occlusion, best corrected visual acuity, cumulative blood vessel length, and corneal neovascularization area.

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinically stable corneal neovascularization who were not improved after treatment with 1% prednisolone acetate eyedrops instilled 4 times a day for at least 1 month

Exclusion Criteria:

* Individuals who had active keratitis with vessel proliferation, uncontrolled inflammation, active hepatitis or clinically significant liver disease, or porphyria or other porphyrin sensitivity

Ages: 35 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Kyung chul Yoon, MD, Study Director — Chonnam natianl university hospital